CLINICAL TRIAL: NCT03916861
Title: Bioelectrical Impedance Analysis Versus Physician Adjustment in Acute Kidney Injury Patients Requiring Renal Replacement Therapy;Which One Can Help Reduce Intradialytic Hypotension
Brief Title: BIA Versus Physician Adjustment in Acute Kidney Injury Patients Requiring Renal Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Responsible Party: Principal Investigator, Thananda Trakarnvanich, Associate Professor, Bangkok Metropolitan Administration Medical College and Vajira Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106/60
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Intradialytic Hypotension; Cardiac Event; Renal Insufficiency; Hospital Length of Stay
Keywords: Hemodialysis; BIA; Acute Kidney Injury
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Intervention Model Description: Prospective randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioelectrical Impedance (Experimental): The first group will be monitored by Inbody S20 analysis to measure fluid status. The Bioimpedance will be measured each time prior to hemodialysis session . The value of BIA measurement of more than 0.4 will be considered as edema.
  Interventions: Device: Bioelectrical Impedance Analysis
- Physicain-guided group (Active Comparator): The fluid monitoring will be managed by physician-adjustment by physical examination and fluid balance record . The fluid balance (FB) is the total fluid administered minus the total fluids eliminated over a period of time.
  Interventions: Procedure: Physician-guided

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis — We use Inbody S20 analysis to measure fluid status before each hemodialysis session to guide fluid removal.
  Arms: Bioelectrical Impedance
Procedure: Physician-guided — This intervention used physical examination as guided to adjust fluid therapy together with the chart record of intake and output per day
  Other Names: Fluid balance record
  Arms: Physicain-guided group

SUMMARY:
This study was designed to compare the efficacy of BIA and physician adjustment to prevent intradialytic hypotension in patients with acute kidney injury who received renal replacement therapy. The investigators randomized 9 patients with acute kidney injury and volume overloaded who underwent acute hemodialysis for 45 sessions in Vajira hospital between October 2017 and February 2018. In physician adjust-group (control) estimate by physical examination and fluid balance record. Primary outcome was intradialytic hypotensive episode and secondary outcome was hemodialysis-related adverse events and other clinical outcome.

DETAILED DESCRIPTION:
Background

Volume overload and intradialytic hypotension are significant complications with increasing mortality rate in hemodialysis patients. Bioelectrical Impedance Analysis (BIA) has been used to estimate the optimum weight in chronic hemodialysis patient to prevent intradialytic hypotension.Volume assessment in acute kidney injury is also of great importance , however, there are currently few methods to obtain an accurate assessment of hydration status in this scenario. This study was designed to compare the efficacy of BIA and physician adjustment to prevent intradialytic hypotension in patients with acute kidney injury who received renal replacement therapy.

Methods

The investigators randomized 9 patients with acute kidney injury and volume overloaded who underwent acute hemodialysis for 45 sessions in Vajira hospital between October 2017 and February 2018. Volume overload was defined by BIA with value more than>0.4. In physician adjust-group (control) estimate by physical examination and fluid balance record. Primary outcome was intradialytic hypotensive episode and secondary outcome was hemodialysis-related adverse events and other clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute kidney injury with volume overload unresponsive to medication therapy =Required renal replacement therapy (RRT)

Exclusion Criteria:

Patients who were pregnant

* Advanced malignancy
* Kidney transplantation
* AKI from toxins
* Currently on pacemaker
* Had underlying chronic kidney disease
* Patients with severe cardiovascular disease such as congestive heart failure, valvular regurgition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — More than 18 years old
Enrollment: 9 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure during dialysis | During hemodialysis session start from enrollment until study completion, up to 4 hours
  Blood pressure less than 20 mmHg from baseline ( systolic blood pressure)

SECONDARY OUTCOMES:
Cardiac problem | Measure through study completion,for at least 3 months after randomization
  Number of patients that have palpitation,cardiac arrthymia or chest pain
Hospital length of stay | Up to 3 months after enrollment
  Total days in admission
Percent of renal function | at least 3 months after enrollment
  eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Thananda Trakarnvanich, Principal Investigator — Vajira Hospital ,Navamindradhiraj University
Locations (1):
- Thananda Trakarnvanich, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No